CLINICAL TRIAL: NCT02583542
Title: A Phase Ib/IIa Study of AZD2014 in Combination With Selumetinib in Patients With Advanced Cancers
Brief Title: A Study of AZD2014 in Combination With Selumetinib in Patients With Advanced Cancers
Acronym: TORCMEK
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen Mary University of London (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009896QM; 2014-002613-31 (EudraCT Number)
Record Dates: First submitted 2015-01-23; First posted 2015-10-22 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Triple-Negative Breast Cancer; Squamous Cell Lung Cancer; Non-squamous Cell Lung Cancer With KRAS Mutations; Non-squamous Cell Lung Cancer With Wild-type KRAS
Keywords: breast; lung; squamous; KRAS; AZD; selumetinib
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — vistusertib; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Escalation Phase (Phase Ib) (Experimental): This phase will investigate two different dosing schedules of AZD2014: a continuous daily schedule (CC-Schedule) and an intermittent schedule of 2 days on and 5 days off treatment (IC-Schedule). The dose of Selumetinib (AZD6244) will remain unchanged in both schedules. The outcome of this investigation will determine whether an additional schedule of combined intermittent Selumetinib (AZD6244) (3 days on and 4 days off treatment) with intermittent AZD2014 will be considered (II-Schedule). The II-Schedule will be initiated following the completion of the corresponding continuous regimens and will only be investigated if escalation of the AZD2014 dose in the IC-Schedule is not feasible with the corresponding continuous Selumetinib (AZD6244) regimen. Up to three individual dose levels of Selumetinib (AZD6244) might subsequently be explored within the intermittent schedule of Selumetinib (AZD6244).
  Interventions: Drug: AZD2014; Drug: AZD6244
- Dose Expansion Phase (Phase IIa) (Experimental): Following the definition of the recommended Phase 2 Dose (RP2D), three NSCLC and one TNBC dose expansion cohorts are planned to perform a preliminary assessment of the anti-tumour efficacy in different molecular settings and to further establish the safety profile of the selected RP2D. These cohorts are:
  * Triple-negative breast cancer (TNBC)
  * Squamous cell lung cancers
  * Non-squamous cell lung cancers with KRAS mutations
  * Non-squamous cell lung cancers with wild-type KRAS
  Interventions: Drug: AZD2014; Drug: AZD6244

INTERVENTIONS:
Drug: AZD2014 — AZD2014 is a dual inhibitor of both mTORC1 (rapamycin-sensitive) and mTORC2 (rapamycin insensitive); compared to rapalogues, AZD2014 has a broader range of growth inhibitory activity in preclinical models based on a more profound mTORC1 inhibition and the additional inhibition of mTORC2. AZD2014 is currently in phase 2 studies in renal cell cancers and metastatic breast cancer.
Drug: AZD6244 — Selumetinib (AZD6244, ARRY-142886) is an orally available, potent, selective, non-ATP competitive inhibitor of MEK1/MEK2 kinases. Selumetinib has demonstrated clinical efficacy in pre-treated KRAS-mutant NSCLC, leading to a significantly improved progression-free survival in combination with docetaxel compared to docetaxel alone.
  Other Names: Selumetinib

SUMMARY:
Open-label, multicentre phase Ib/IIa study of AZD2014 administered with selumetinib. There are two parts to this study: a dose-escalation part in treatment-refractory advanced solid tumours and a subsequent separate expansion cohort part for TNBC, squamous cell lung cancers, non-squamous cell lung cancers with KRAS mutations and non-squamous cell lung cancers with wild-type KRAS

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to admission to this study
2. Age ≥18 years
3. ECOG performance status 0 or 1
4. Life expectancy ≥12 weeks
5. Patients must have at least one lesion, not previously irradiated, that can be measured accurately at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements
6. Radiological or clinical evidence of disease progression
7. Formalin fixed, paraffin embedded tumour sample from the primary or recurrent cancer must be available for central testing
8. Adequate haematologic and end organ function, defined by the following laboratory results obtained within 7 days prior to the first study treatment:

   * ANC ≥ 1.5 x 109/l (without granulocyte colony-stimulating factor support within 2 weeks prior to the first study treatment)
   * Platelet count ≥ 100 x 109/l (without transfusion within 2 weeks prior to the first study treatment)
   * Haemoglobin ≥ 9 g/dl (transfusion permitted to establish target haemoglobin levels prior to the first study treatment)
   * Serum creatinine ≤1.5 times the upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 ml/min
   * Bilirubin level ≤1.5 x ULN (patients with known Gilbert disease who have bilirubin levels ≤ 3 x ULN may be enrolled)
   * AST or ALT <2.5 x ULN or <5 x ULN in the presence of liver metastases
   * Alkaline phosphatase (ALP) <2.5 x ULN or <5 x ULN in the presence of liver and/or bone metastases
   * INR and aPTT ≤1.5 x ULN; this applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
   * Female patients of child-bearing potential are eligible, provided they have a negative serum or urine pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible. All patients with reproductive potential must agree to use adequate contraception beginning two weeks before the first dose of investigational product and for three months after the discontinuation of treatment. Adequate contraception methods include: intrauterine device [IUD], birth control pills unless clinically contraindicated, or a barrier device.

Inclusion Criteria unique to the Dose Escalation Part (phase Ib part):

1. Histologically or cytologically advanced solid tumour limited to:

   * Tumour types with frequent activation of MAPK and/or PI3K pathways (pancreatic, thyroid, endometrial, renal, breast or ovarian carcinoma, colorectal cancer, NSCLC or melanoma) OR
   * Tumours with known alteration in ≥1 gene involved in PI3K/AKT/mTOR or Ras/MEK pathway signalling, such as: KRAS, NRAS, BRAF, PIK3CA, PTEN, AKT, LKB1, EGFR, FGFR, HER2, MET, RET, KIT, NF1
2. Metastatic or locally advanced disease, which is refractory to conventional treatment or for which no conventional therapy exists; locally recurrent disease must not be amenable to resection with curative intent (patients who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible).

Inclusion Criteria unique to the lung cancer dose expansion cohorts (phase IIa part):

1. Histologically confirmed NSCLC
2. Stage III disease that is unsuitable to radio-chemotherapy or Stage IV disease or recurrent NSCLC; recurrent disease must not be amenable to resection or radical radiotherapy with curative intent.
3. Prior chemotherapy and/or, if indicated/accessible, EGFR-directed or ALK-directed therapy for advanced disease

Inclusion Criteria unique to the TNBC dose expansion cohort (Phase IIa):

1. Histologically confirmed TNCB defined as tumour cells being:

   * Negative for ER with <1% of tumour cells positive for ER on IHC or IHC score (Allred) of ≤2
   * Negative for PR with <1% of tumour cells positive for PR on IHC or IHC score (Allred) of ≤2 or PR unknown, and
   * Negative for HER2 with 0, 1+ or 2+ intensity on IHC and no evidence of amplification on ISH.
2. Metastatic or locally recurrent disease; locally recurrent disease must not be amenable to resection with curative intent (patients who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible).
3. Prior chemotherapy for advanced disease

Exclusion Criteria:

1. Symptomatic CNS involvement or CNS involvement requiring steroid therapy; patients with treated brain metastases that are asymptomatic and have been clinically stable for 1 month will be eligible for protocol participation
2. Prior chemotherapy, biological therapy, radiation therapy, immunotherapy, other anticancer agents and any investigational agents within 14 days of starting study treatment (not including palliative radiotherapy at focal sites)
3. Any unresolved toxicity > CTCAE Grade 1 from previous anti-cancer therapy, with the exception of alopecia
4. Current refractory nausea and vomiting, chronic gastrointestinal disease or inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of the study medication
5. Significant cardiovascular disease, such as;

   * History of myocardial infarction, acute coronary syndromes (including unstable angina), or coronary angioplasty/stenting/bypass grafting within past 6 months.
   * Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy)
   * History of symptomatic congestive heart failure (CHF) New York Heart Association (NYHA) Classes II-IV or Left ventricular ejection fraction (LVEF) <55% measured by echocardiography
   * Severe cardiac arrhythmia requiring medication or severe conduction abnormalities (unless compensated by ventricular pacemaker); atrial fibrillation with a ventricular rate >100 bpm on ECG at rest
   * Poorly controlled hypertension (resting diastolic blood pressure >115 mmHg)
   * Clinically significant valvular disease, cardiomegaly, ventricular hypertrophy, or prior or current cardiomyopathy
6. QTc prolongation defined as a QTc interval >470 msecs
7. Concomitant medications known to prolong QT interval
8. Patients receiving concomitant immunosuppressive agents or chronic systemic corticosteroids (≥ 10 mg prednisolone or an equivalent dose of other anti-inflammatory corticosteroids) use for ≥ 28 days at the time of study entry except in cases outlined below: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed. Patients on stable low dose (<10 mg prednisolone or an equivalent dose of other anti-inflammatory corticosteroids) of corticosteroids for at least two weeks before registration are allowed
9. Evidence of interstitial fibrotic lung disease (bilateral, diffuse, parenchymal lung disease)
10. Clinically significant abnormalities of glucose metabolism as defined by any of the following

    * Diagnosis of diabetes mellitus type I or II (irrespective of management).
    * Glycosylated haemoglobin (HbA1C) ≥ 8.0% at screening (64 mmol/mol) (conversion equation for HbA1C [IFCC-HbA1C (mmol/mol) = [DCCT-HbA1C (%) - 2.15] x 10.929)
    * Fasting Plasma Glucose ≥ 7.0mmol/L (126 mg/dL) at screening. Fasting is defined as no caloric intake for at least 8 hours.
11. Ophthalmological conditions as follows:

    * Intra-ocular pressure >21 mmHg, or uncontrolled glaucoma (irrespective of intra-ocular pressure)
    * Current or past history of central serous retinopathy or retinal vein occlusion
12. Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 if taken within the stated washout periods before the first dose of study treatment

    * Inhibitors (competitive): ketoconazole, itraconazole, indinavir, saquinovir, nelfinavir, atazanavir, amprenavir, fosamprenavir, troleandomycin, telithromycin, fluconazole, nefazodone, cimetidine, aprepitant, miconazole, fluvoxamine, P-glycoprotein, grapefruit juice, or seville oranges (1 week minimum wash-out period), amiodarone (27 week minimum wash-out period)
    * Inhibitors (time dependent): erythromycin, clarithromycin, verapamil, ritonavir, diltiazem (2 week minimum wash-out period)
    * Inducers: phenytoin, rifampicin, St. John's Wort, carbamazepine, dexamethasone, primidone, griseofulvin, carbamazepine, barbiturates, troglitazone, pioglitazone, oxcarbazepine, nevirapine, efavirenz, rifabutin (3 week minimum wash-out period) and phenobarbitone (5 week minimum wash-out period)
13. Exposure to potent or moderate inhibitors or inducers of CYP2C8 within the stated washout periods before the first dose of study treatment

    * Inhibitors: Gemfibrozil, trimethoprim, glitazones, montelukast, quercetin (1 week minimum wash-out period)
    * Inducers: Rifampicin (3 week minimum wash-out period)
14. Exposure to sensitive or narrow therapeutic range substrates of the drug metabolising enzymes CYP2C8, CYP2C9, CYP2C19, CYP2D6 or the drug transporters Pgp (MDR1) and BCRP within the appropriate wash-out period before the first dose of study treatment
15. Active second malignancy (except non-melanomatous skin cancer): active secondary malignancy is defined as a current need for cancer therapy or a high possibility (>30%) of recurrence during the study.
16. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
17. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
18. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.
19. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug ≤30 days prior to study entry depending on the half-life of the investigational drug and/or guidance issued by the TORCMEK IMP manufacturer. Please contact the TORCMEK Coordinating team for further information.

Exclusion Criteria unique to the dose expansion cohorts (phase IIa part):

1. Prior treatment with PI3K inhibitors, AKT inhibitors, mTOR inhibitors or MEK, Ras or Raf inhibitors.
2. Prior radiotherapy to the indicator lesion(s); Newly arising lesions in previously irradiated areas are accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2015-06; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Establish feasible dose levels and regimens of AZD2014 and selumetinib when given in combination by close observation of any dose limiting toxicities | First 21 days of treatment.
  Dose limiting toxicity is defined as occurrence of any of the following toxicities during the first 21 days of treatment:
  * Any grade >3 non-haematological toxicity (excluding nausea, vomiting or diarrhoea)
  * Grade 3 nausea, vomiting or diarrhoea lasting >48 hours despite supportive care or any Grade 4 hause, vomiting or diarrhoea
  * Grade 4 neutropenia lasting >7days or febrile neutropenia
  * Grade 3 thrombocytopenia with bleeding or grade 4 thrombocytopenia
  * Inability to receive at least 75% of the planned doses due to unresolved toxicity
  * Any treatment delays for >14 days due to unresolved toxicity
  NB: This primary outcome relates to the Phase Ib part of study.
Assess clinical activity, as measured by disease control rate, of AZD2014 in combination with selumetinib. | Day 1 to > 12 weeks.
  Disease control rate is defined as number of patients with complete or partial response or stable disease maintained >12weeks (as assessed by the site radiologist and/or investigator, using RECIST 1.1) divided by the number of patients in the analysis. Patients without a post-baseline tumour assessment will be considered to have no disease control.
  NB: This primary outcome relates only to the Phase IIa part of this study

SECONDARY OUTCOMES:
Single dose and/or multiple dose AZD2014 PK Tmax parameters will be used to determine the PK of AZD2014 when given in combination with selumetinib. | Until Day 9
Single dose and/or multiple dose AZD2014 PK Cmax parameter will be used to determine the PK of AZD2014 when given in combination with selumetinib. | Until Day 9
Single dose and/or multiple dose AZD2014 PK AUC parameters will be used to determine the PK of AZD2014 when given in combination with selumetinib. | Until Day 9
Assess clinical activity of AZD2014 and Selumetinib, as measured by objective response rate. | 12 weeks.
  Objective response, defined as a complete or partial response (as assessed by the site radiologist and/or investigator, using RECIST 1.1) divided by the number of patients of risk
Assess clinical activity of AZD2014 and Selumetinib, as measured by change in tumour size. | 12 weeks.
  Average change (%) in tumour size at 12 weeks compared to baseline, as assessed by RECIST 1.1; tumour size is defined as the sum of the diameters of the target lesion.
To assess the safety and tolerability of AZD2014 when given in combination with selumetinib by the continuous assessment of Adverse Events. | A median time of 12 weeks.
  i.e. Incidence of serious adverse events; Incidence of Grade 3 and 4 adverse events; Incidence of all adverse events of all grades; Adverse events leading to discontinuation of the study medication; Clinically significant changes in vital signs and clinical laboratory results during and following study drug administration; Clinically significant changes in ECG measurements
Overall survival defined as the time from date of registration to the date of death due to any cause will be used to assess the efficacy of AZD2014 when given in combination with selumetinib. | A median time of 12 weeks.
Duration of response will be used to assess of AZD2014 when given in combination with selumetinib. | A median time of 12 weeks.
  Duration of response defined as the time from first documentation of CR or PR to disease progression (RECIST v1.1) or death from any cause, whichever occurs first.
Single dose and/or multiple dose of AZD2014 and selumetinib PK Tmax parameters will be used to investigate the PK of Selumetinib when given in combination with AZD2014. | Until Day 9
Single dose and/or multiple dose of AZD2014 and selumetinib PK Cmax parameters will be used to investigate the PK of Selumetinib when given in combination with AZD2014. | Until Day 9
Single dose and/or multiple dose of AZD2014 and selumetinib PK AUC parameters will be used to investigate the PK of Selumetinib when given in combination with AZD2014. | Until Day 9
Progression-free survival (PFS) will be used to assess the efficacy of AZD2014 when given in combination with selumetinib. | A median time of 12 weeks.
  PFS defined as the time from the date of registration to the date of first documented tumour progression (RECISTv1.1) or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Professor, Study Director — Queen Mary University
Locations (4):
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Christie NHS Foundation Trust, Manchester